CLINICAL TRIAL: NCT01699477
Title: MR-Guided Functional Ultrasound-Neurosurgery
Brief Title: Safety Study Using Transcranial MR Guided Focused Ultrasound in the Treatment of Neuropathic Pain
Acronym: FUS-CLT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: E-04/2008
Record Dates: First submitted 2012-04-27; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Functional Brain Disorders /Neuropathic Pain
Keywords: FUS; focused ultrasound; functional brain disorders; neuropathic pain; movement disorders
MeSH Terms: conditions — Neuralgia; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trancranial MRg Focused Ultrasound for Neuropatic Pain (Other)
  Interventions: Device: ExAblate 4000 focused ultrasound brain intervention

INTERVENTIONS:
Device: ExAblate 4000 focused ultrasound brain intervention — Non-invasive brain intervention using MR-guided focused ultrasound

SUMMARY:
The aim of this study is to asses the efficacy and the clinical safety of the transcranial magnetic resonance guided high intensity focused ultrasound system ExAblate 4000, InSightec Ltd. for functional neurosurgery. The treatments to be conducted in this study are non-invasive, i.e. without opening the skull, and will create micro-thalamotomies in specific target areas such as thalamus, subthalamus and pallidum. The data obtained in this study will be used to evaluate the basic safety aspects of this new treatment technology and will serve as a basis for the clinical introduction of MR-guided ultrasound-neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years and older
2. Clinical indication for a medial thalamotomy
3. Stereotactic targets within thalamus, subthalamus and pallidum
4. All targets supposedly accessible by TcMRgFUS
5. Physically and mentally able to understand the risks of participating in this study and to give written informed consent based on the patient information provided
6. Sufficient proficiency in one of the languages German, French, Italian or English to al-low for verbal communication during all phases of the study
7. Physically and mentally able to communicate the personal condition and all feelings during the TcMRgFUS treatment
8. Physically and mentally able to undergo the TcMRgFUS treatment

Exclusion Criteria:

1. Anomalies of brain anatomy, especially in or around thalamus or pallidum that will in-fluence the atlas-based navigation
2. Existing lesions in close proximity (<5mm) to planned ablation targets
3. Extended anomalies of scalp such as scars, inflammations, etc.
4. Clips or other implanted objects close to (< 3cm) target
5. Non-MRI-compatible cardiac pacemaker
6. Previous hemorrhages in the brain
7. Uncontrolled arterial hypertension
8. Any coagulopathy or patient under anticoagulant therapy
9. Sensitivity to MRI contrast agents
10. Contraindications to MRI such as non-MRI-compatible implanted devices
11. Large patients not fitting comfortably into the MRI unit (generally >110kg)
12. Difficulty to lie supine and still for up to 4 hours in the MRI unit or claustrophobia
13. Other known life-threatening systemic disease
14. Patients currently participating or participated in another clinical trial in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Precision of lesioning | 3 months
  Comparison of size and location of sonicaion lesions on MRI with planning coordinates.
Safety measurements | 6 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability.
Lesion characteristics | 3 months
  Size of lesions as a function of applied energy/temperature.

SECONDARY OUTCOMES:
Clinical Efficacy | 1 year
  Pain Scores on the Visual Analog Scale following intervention and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst - Martin, MD, Principal Investigator — University Children's Hospital, Zurich; Ronald - Bauer, MD, Principal Investigator — Neurosurgery, Kantonsspital St. Gallen, Switzerland; Gunther - Landmann, MD, Principal Investigator — Center for Pain Medicine, Nottwil, Switzerland
Locations (1):
- MR-Center, University Children's Hospital, Zurich, Canton of Zurich, Switzerland